CLINICAL TRIAL: NCT05387551
Title: Effect of Adding Continuous Glucose Monitoring (CGM) to Lifestyle Changes on Insulin Sensitivity in Patients With Impaired Glucose Tolerance
Brief Title: CGM and Lifestyle Changes in Patients With Impaired Glucose Tolerance
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nemours Children's Clinic (Other)
Responsible Party: Principal Investigator, Larry A. Fox, MD, Division Chief, Nemours Children's Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: lfox051622
Record Dates: First submitted 2022-05-16; First posted 2022-05-24 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Impaired Glucose Tolerance; Prediabetes
Keywords: impaired glucose tolerance; obesity; adolescents
MeSH Terms: conditions — Glucose Intolerance; Prediabetic State; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- CGM intervention (Experimental): Continuous glucose monitoring with real-time glucose data using Dexcom G6.
  Interventions: Device: CGM

INTERVENTIONS:
Device: CGM — Dexcom G7 sensor, transmitter and supplies will be provided to family for use. Participants will wear G7 and have real-time glucose data throughout the study.
  Other Names: Dexcom G7

SUMMARY:
The incidence of type 2 diabetes (T2D) in children is increasing, paralleling the rising incidence of obesity. Preventing children and adolescents from developing T2D is critical. The health benefits of lifestyle modifications are well documented in this population, but success rates are low. Obesity in children and adolescents increases the risk of not only T2D but other complications as well, such as hypertension, dyslipidemias and more. The investigators hypothesize that having real-time glucose data with the use of a continuous glucose monitor (CGM) in obese patients with impaired glucose tolerance will improve adherence to lifestyle modifications. As a result, a decrease in body mass index (BMI) is expected with subsequent improvement in insulin sensitivity, thus reducing risk of obesity-related complications later in childhood/adolescence and adulthood.

DETAILED DESCRIPTION:
The purpose of this research is to evaluate if having blood sugar information from a continuous glucose monitor (CGM) during activities of daily living provides additional benefit to lifestyle modifications in reducing the risk of developing diabetes and achieving a healthier weight. A CGM is a small device often worn on the back of the arm that uses a very small needle to insert a small sensor just under the skin in the fatty tissue. The CGM device transmits the blood sugar level to either a smartphone or a special receiver.

The investigators expect patients will have an overall improvement in health by decreasing weight and therefore improving the way the child's insulin works in their body. This could result in decreased risk of obesity-related complications such as diabetes mellitus, cardiovascular disease, kidney disease, and loss of vision and/or limbs, among others.

ELIGIBILITY:
Inclusion Criteria:

1. Children 10 to <18 years old (i.e., before their 18th birthday)
2. Impaired glucose tolerance based on standardized oral glucose tolerance test (OGTT) or fasting glucose per American Diabetes Association criteria,
3. Overweight or obese (BMI ≥85th percentile for age/sex)
4. Patients are pubertal, defined as females with breast Tanner stage II or above, or males with testicular volume ≥4 mL

Exclusion Criteria:

1. Existing diagnosis of type 1 or type 2 diabetes
2. Prepubertal
3. Taking medications that affect insulin sensitivity (e.g.,chronic corticosteroids whether systemic or inhaled). Metformin allowed if stable dose.
4. Patients and/or families not willing to wear the CGM for the duration of the study period or lack of compliance after recruitment

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Insulin Sensitivity Score (ISS) | Baseline to 6 months
  Change in insulin sensitivity as measured by insulin sensitivity Score (ISS). The ISS directly correlates with insulin sensitivity. Higher scores indicate higher insulin sensitivity; lower scores indicate more insulin resistance.

SECONDARY OUTCOMES:
QUICKI insulin sensitivity | Baseline to 3 months
  Change in insulin sensitivity as measured by QUICKI
QUICKI insulin sensitivity | Baseline to 6 months
  Change in insulin sensitivity as measured by QUICKI
Insulin Sensitivity Score | Baseline to 3 months
  Change in insulin sensitivity as measured by insulin sensitivity Score (ISS). The ISS directly correlates with insulin sensitivity. Higher scores indicate higher insulin sensitivity; lower scores indicate more insulin resistance.
Glycemic levels | Baseline to 3 and 6 months
  Change in characteristics of glycemic levels obtained from the CGM data. This will include:
  * mean, standard deviation of glucose levels
  * time in range (glucose between 70-140 mg/dL)
  * percent of time with hyperglycemia (>140 mg/dL)
  * percent of time with hypoglycemia (<70 mg/dL)
Mean, standard deviation of sensor glucose levels | Baseline to 3 and 6 months
  Change in characteristics of glycemic levels obtained from the CGM data, including mean and standard deviation of sensor glucose levels (mg/dL).
Time in range of sensor glucose levels | Baseline to 3 and 6 months
  Change in glycemic levels obtained from the CGM data: Percent of time in range (glucose between 70-140 mg/dL)
Percent of sensor glucose levels in hypoglycemic range | Baseline to 3 and 6 months
  Change in glycemic levels obtained from the CGM data: Percent of time with hypoglycemia (<70 mg/dL)
Percent of sensor glucose levels in hyperglycemic range | Baseline to 3 and 6 months
  Change in glycemic levels obtained from the CGM data: Percent of time with hyperglycemia (>140 mg/dL)
Physical activity questionnaires | 3 and 6 months
  Questionnaires will be used to assess amount of time participants are active. Two questions regarding physical activity will be asked, with a scale set up as follows:
  1. How many minutes of continuous physical activity per week were completed? Possible answers will be <10, 11-20, 21-30, 31-60, 61-90, 91-120, or 121-150.
  2. How many days per week of physical activity longer than 30 minutes? Possible answers will be 0, 1, 2, 3, 4, 5, 6, or 7.
Dietary compliance questionnaires | 3 and 6 months
  Questionnaires will be used to assess particpants' compliance witih dietary changes. Four questions regarding their diet will be asked, with a scale set up as follows:
  1. How many sugary drinks per week? Possible answers will be 0, 1-2, 3-5, or >5.
  2. How many unhealthy snacks per week? Possible answers will be 0, 1-2, 3-5, or >5.
  3. How many times junk food was consume in the past week? Possible answers will be 0, 1-2, 3-5, or >5.
  4. How often were the proper portion sizes followed (as per control plate)? Possible answers will be always, most days, occasionally, or never.

CONTACTS AND LOCATIONS:
Overall Officials: Larry A Fox, MD, Principal Investigator — Nemours Children's Health
Locations (1):
- Nemours Children's Clinic, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No